CLINICAL TRIAL: NCT05525442
Title: Factors Affecting The Recurrence Of Acute Cholecystitis After Treatment With Percutaneous Cholecystostomy
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Korhan TUNCER, General Surgeon, Tepecik Training and Research Hospital
Other Study IDs: 2021/05-12
Record Dates: First submitted 2022-07-16; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Acute Cholecystitis; Percutaneous Cholecystostomy; Recurrence
Keywords: acute cholecystitis; percutaneous cholecystostomy; Tokyo guidelines 2018; recurrence
MeSH Terms: conditions — Cholecystitis, Acute; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with recurrence: Recurrence in the first year after percutaneous cholecystostomy catheter removal
  Interventions: Procedure: percutaneous cholecystostomy
- patients without recurrence: No recurrence within the first year after percutaneous cholecystostomy catheter removal
  Interventions: Procedure: percutaneous cholecystostomy

INTERVENTIONS:
Procedure: percutaneous cholecystostomy — Transhepatic gallbladder drainage was performed under ultrasound guidance after local anesthesia was administered by interventional radiology to patients with acute cholecystitis. Subsequently, an 8-10 Fr pigtail catheter was inserted into the gallbladder using a guide wire under fluoroscopy.

SUMMARY:
Percutaneous cholecystostomy is used to reduce the complications and mortality associated with surgery in patients with high surgical risk in acute cholecystitis. Although this method generally acts as a bridge treatment for interval cholecystectomy in patients, interval cholecystectomy is not performed in every patient after percutaneous cholecystostomy. The aim of this study was to determine the recurrence rate of patients who did not have interval cholecystectomy after treatment with percutaneous cholecystostomy and to investigate the factors that may affect the recurrence.

DETAILED DESCRIPTION:
Acute cholecystitis is an inflammatory disease of the gallbladder and is often associated with cholelithiasis. According to Tokyo Guide 2018 (TG18), acute cholecystitis is grouped with various risk factors and predictive factors. Early laparoscopic cholecystectomy or late cholecystectomy after medical therapy is recommended for patients with grades 1 and 2. On the other hand, non-operative treatments such as percutaneous cholecystostomy catheter and antibiotic therapy are recommended for selected patients with high surgical risk and serious comorbidities in order to prevent morbidity and mortality. They suggested that percutaneous cholecystostomy catheter could be used as the definitive treatment of acute cholecystitis in these high-risk patients who are not suitable for surgery. Debate continues as to whether cholecystectomy is necessary for these patients. Because studies have shown that the recurrence rate of acute cholecystitis after percutaneous cholecystostomy catheter treatment varies between 4% and 22%. For these reasons, assessing the risk of recurrence of acute cholecystitis in patients initially treated with percutaneous cholecystostomy is essential to aid decision making.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute cholecystitis on admission to the emergency department
* Patients treated with percutaneous cholecystostomy catheter according to TK18 acute cholecystitis diagnosis and treatment guideline
* Patients older than 18 years
* Patients who can give their own consent

Exclusion Criteria:

* Patients with missing data or not followed up regularly
* Patients whose cholecystostomy catheter was removed during the operation or operated within the first year following the catheter extraction
* Patients with choledocholithiasis, abscess secondary to acute cholecystitis, or hepatopancreatobiliary system malignancy
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with percutaneous cholecystostomy catheter due to acute cholecystitis will be included in the study. Admission to hospital up to 1 year after the acute cholecystitis attack will be retrospectively screened through the hospital data system. The collected data will be statistically analyzed in SPSS.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
recurrence | one year
  Factors affecting recurrence will be investigated in patients who underwent percutaneous cholecystostomy catheter for acute cholecystitis. These factors; age, gender, comorbidities, presence of fever, history of previous cholecystitis attack, catheter insertion time, catheter drainage time, reproduction in bile culture, gallbladder content, various laboratory parameters, gallbladder wall thickness and diameter, Tokyo classification vs.

CONTACTS AND LOCATIONS:
Overall Officials: Korhan Tuncer, MD, Principal Investigator — Tepecik Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Kiriyama S, Kozaka K, Takada T, Strasberg SM, Pitt HA, Gabata T, Hata J, Liau KH, Miura F, Horiguchi A, Liu KH, Su CH, Wada K, Jagannath P, Itoi T, Gouma DJ, Mori Y, Mukai S, Gimenez ME, Huang WS, Kim MH, Okamoto K, Belli G, Dervenis C, Chan ACW, Lau WY, Endo I, Gomi H, Yoshida M, Mayumi T, Baron TH, de Santibanes E, Teoh AYB, Hwang TL, Ker CG, Chen MF, Han HS, Yoon YS, Choi IS, Yoon DS, Higuchi R, Kitano S, Inomata M, Deziel DJ, Jonas E, Hirata K, Sumiyama Y, Inui K, Yamamoto M. Tokyo Guidelines 2018: diagnostic criteria and severity grading of acute cholangitis (with videos). J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):17-30. doi: 10.1002/jhbp.512. Epub 2018 Jan 5. PMID 29032610
- [Result] Leveau P, Andersson E, Carlgren I, Willner J, Andersson R. Percutaneous cholecystostomy: a bridge to surgery or definite management of acute cholecystitis in high-risk patients? Scand J Gastroenterol. 2008;43(5):593-6. doi: 10.1080/00365520701851673. PMID 18415753
- [Result] Sanjay P, Mittapalli D, Marioud A, White RD, Ram R, Alijani A. Clinical outcomes of a percutaneous cholecystostomy for acute cholecystitis: a multicentre analysis. HPB (Oxford). 2013 Jul;15(7):511-6. doi: 10.1111/j.1477-2574.2012.00610.x. Epub 2012 Nov 19. PMID 23750493
- [Result] Li M, Li N, Ji W, Quan Z, Wan X, Wu X, Li J. Percutaneous cholecystostomy is a definitive treatment for acute cholecystitis in elderly high-risk patients. Am Surg. 2013 May;79(5):524-7. doi: 10.1177/000313481307900529. PMID 23635589